CLINICAL TRIAL: NCT04265859
Title: Changes in Brain Function Through Repeated Emotion Regulation Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Stevens (Other)
Responsible Party: Sponsor-Investigator, Michael Stevens, Senior Research Scientist, Hartford Hospital
Organization: Hartford Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-HCC-2016-0177
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Adults having mild-to-moderate levels of depression or who will serve as non-depressed/anxious controls. Participants in each of these study groups then will be randomized into two conditions, each of which will receive 2 assessment/MRI appointments along with 6 sessions of guided practice/training in either 1) Re-interpretation or 2) Mindfulness ER techniques. Immediately after the first and sixth practice sessions, participants also will undergo fMRI so that brain function relative to that stage of practice can be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depressed (Experimental): Participants in this group will be randomized to receive either the CBT training (n=10) or Mindfulness training (n=10).
  Interventions: Behavioral: Cognitive Behavioral Training; Behavioral: Mindfulness
- Healthy Control (Other): Participants in this group will be randomized to receive either the CBT training (n=10) or Mindfulness training (n=10).
  Interventions: Behavioral: Cognitive Behavioral Training; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Cognitive Behavioral Training — The CBT-based regulation training involves using a cognitive strategy that instructs participants to reappraise situations in positive or less negative ways.
  Other Names: CBT
Behavioral: Mindfulness — The MBT-based regulation training involves using a mindfulness strategy that instructs participants to notice and accept their feelings without judgment or intent to act upon them.

SUMMARY:
This is a pilot study that will investigate how two psychotherapies (re-interpretation and mindfulness) alter brain function. This information will be used to gain understanding of how repeated emotion regulation practices influence the brain and to develop a focused, tactic-based emotional regulation remediation approach for treatment of ADHD.

DETAILED DESCRIPTION:
The goal of this pilot study is to collect preliminary data that will allow the investigators to formulate theories about ER-related brain function change during intervention-like training that will be tested in larger, externally-funded grant proposals submitted to the National Institutes of Health. The investigators are not especially interested in any existing specific, manualized therapeutic technique. Existing ER-based psychotherapies typically incorporate a variety of related interventions, not all of which focus on the ER component itself. Instead, the investigators will focus on the "building blocks" of such therapies, i.e., the ER interventions themselves and their effect on negative emotional reactions. Here, the investigators ask a specific question - How does ER-elicited brain function change with repeated sessions of guided practice of various ER techniques? In other words, does increasing familiarity or mastery of ER skills through practice change brain function, and how? There are logical hypotheses about the likely nature of brain function changes that can be gleaned from prior neuroimaging research. For instance, if prefrontal cortex activation is important to ER, perhaps practice simply increases such activation. However, pilot work for the current NIMH R01 suggests instead that ER practice might work by enhancing the functional integration among key frontolimbic regions. Complicating such hypotheses is the recognition that different ER tactics engage many distinct brain regions depending on which approach is employed. So a participant's individual brain function differences prior to ER training might be a potent determinant for what sorts of neural changes result from repeated practice. Because all these issues must be evaluated through the lens of a preliminary study before any coherent theoretical model can be formulated, a pilot study is proposed here. Not only will this provide empirical data upon which to base future research, conducting such a pilot will showcase any methodological hurdles or challenges that need to be overcome in order to successfully conduct a larger-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Right-handed
* High-school level of education (11th grade attainment for 18 year-olds is acceptable if they haven't completed their final year yet)
* >8th grade English reading level to complete self-report evaluations (most are only available in English).
* For the depressed group, elevated scores on the Beck Depression Inventory - II to validate depressive symptoms.

Exclusion Criteria:

* Head injury sufficient to have caused >30 minutes lost consciousness
* Past or current CNS disease (e.g., MS, epilepsy, tumor, etc.)
* Brain lesion identified by MR (structural MR scans will be reviewed by a radiologist for the presence of clinical neuropathology that may affect cognitive task performance)
* Hypertension or juvenile-onset diabetes (current treatment with antihypertensives or insulin)
* Current pregnancy (menstruating females will be tested)
* DSM-IV Axis I lifetime history of Bipolar disorder, PTSD, OCD, psychotic disorder, Tourette's disorder, or any Pervasive Developmental Disorder (e.g., Autistic disorder, PDD NOS, etc.)
* For the depressed group, current PTSD
* Current DSM-IV substance dependence, ADHD, Conduct Disorder, MDD
* Any current psychotropic medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
fMRI Brain Scan | Visit one and repeated again at Visit two (approximately 4 weeks later)
  fMRI-assessed brain function data, examined either to detect any changes in activation amplitude ("level of activity") in a priori ER-linked brain regions-of-interest (ROIs) or changes in the degree of functional connectivity among them.

SECONDARY OUTCOMES:
Beck Depression Inventory - II and State Trait Anxiety Inventory | Enrollment and repeated again at Visit two (approximately 4 weeks later)
  Depression and anxiety scales (pre and post scores, as evidenced by a decrease in total scores from each scale)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stevens, PhD, Principal Investigator — Institute of Living/Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT04265859/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04265859/ICF_001.pdf